CLINICAL TRIAL: NCT02681523
Title: ALERT: A Phase II Study of Alternating Eribulin and Hormonal Therapy in Pre-treated ER+ve Breast Cancer.
Acronym: ALERT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow patient recruitment
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C/31/2014; 2014-004112-11 (EudraCT Number)
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Results first posted 2021-02-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): 3 x 3 weekly cycles at the recommended dose of eribulin as the ready to use solution, 1.23 mg/m2, administered intravenously over 2-5 minutes on days 1 and 8 of every 21 day cycle. This will then be followed by 9 weeks of AI treatment, to be followed again by 3 x 3 weekly cycles of eribulin and 9 weeks AI treatment. Patients will remain on treatment for up to 9 months, or until disease progression or unacceptable toxicities, whichever is sooner.
  Interventions: Drug: Eribulin

INTERVENTIONS:
Drug: Eribulin
  Other Names: Halaven

SUMMARY:
A single centre, single arm phase II study of alternating eribulin and hormonal therapy in 12 patients with locally advanced or metastatic breast cancer who have received at least one hormonal therapy and at least one chemotherapy in the metastatic setting.

DETAILED DESCRIPTION:
12 patients with locally advanced or metastatic breast cancer who have received at least one hormonal therapy and at least one chemotherapy in the metastatic setting will be enrolled to receive treatment. Once patients are consented and have completed on study screening, eribulin and Aromatase Inhibitor (AI) treatment will be alternated for up to 9 months, until disease progression or unacceptable toxicities, whichever is sooner. Patients will then attend a safety follow-up visit 4 weeks after completing treatment.

Eribulin (Halaven®) is a non-taxane microtubule dynamics inhibitor. Eribulin inhibits the growth phase of microtubules without affecting the shortening phase and sequesters tubulin into non-productive aggregates. Eribulin exerts its effects via a tubulin-based antimitotic mechanism leading to G2/M cell-cycle block, disruption of mitotic spindles, and, ultimately, apoptotic cell death after prolonged mitotic blockage.

Eribulin is licenced for the treatment of patients with locally advanced or metastatic breast cancer who have previously received at least one chemotherapeutic regimen for the treatment of advanced disease. Prior therapy should have included an anthracycline and a taxane in either the adjuvant or metastatic setting unless patients were not suitable for these treatments.

The aim of this study is to alternate eribulin and aromatase inhibitors, examining whether there may be breakthrough relapse during the AI therapy or on the other hand we can extend the duration that eribulin may be used for. Importantly, blood based biomarkers, the tumour derived fraction of circulating free DNA (cfDNA) termed circulating tumor DNA (ctDNA), and circulating tumour cells will be measured. A major aim of this study is to test whether biomarkers fluctuate between chemotherapy and AI treatment in the setting of advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Written informed consent prior to admission to this study
* 2. Aged 18≥over
* 3. Histologically confirmed ER+ve metastatic breast cancer according to local criteria
* 4. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* 5. Have progressed after at least one hormonal therapy regime and at least one chemotherapy regime for advanced disease
* 6. Patients must have had prior treatment with an anthracycline and a taxane (either sequential or in combination) unless patients were not suitable for these treatments. This treatment can be in the adjuvant setting
* 7. Measurable sites of locally advanced and/or metastatic disease that can be accurately assessed by CT/MRI scan at baseline (RECIST v1.1)¹
* 8. Life expectancy of ≥6 months
* 9. Adequate organ function, as defined by:

  * Haemoglobin (Hb) ≥ 9 g/dL
  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelet count (Plts) ≥ 100 x 109/L
  * White Blood Cell (WBC) ≥ 3.0 x 109/L
  * Serum albumin ≤ 1.5 Upper Limit of Normal (ULN)
  * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 3 x ULN if no demonstrable liver metastases or ≤ 5 x ULN in the presence of liver metastases.
  * Alkaline Phosphatase Level (ALP) ≤ 5 x ULN
  * Total bilirubin ≤ 1.5 x ULN if no demonstrable liver metastases or ≤ 3 x ULN in the presence of liver metastases
  * Creatinine ≤ 1.5 x ULN or creatinine clearance >50ml/min
* 10. Postmenopausal as defined by age >50, no menstruation for >2 years, previous oophorectomy or lab results confirming this status
* 11. Premenopausal if has been subject to ovarian ablation/ suppression at least 3 weeks prior to commencing AI therapy

  * RECIST v1.1 updated and now considers bone metastasis with an identifiable soft tissue mass to be measurable disease. Therefore, patients with bone metastasis are eligible, provided they have evaluable disease.

Exclusion Criteria:

* 1.Triple negative or Human Epidermal Growth Factor Receptor 2 (HER2) positive cancer
* 2. Hypersensitivity to the active substance or to any of its excipients
* 3. History of another primary malignancy within 5 years prior to starting study treatment, except adequately treated basal or squamous cell carcinoma of the skin, carcinoma in site and the disease under study
* 4. Evidence of uncontrolled active infection
* 5. Severe hepatic impairment (Child-Pugh C)
* 6. Evidence of significant medical condition or laboratory finding which, in the opinion of the Investigator, makes it undesirable for the patient to participate in the trial
* 7. Concurrent therapy with any other investigational agent or everolimus
* 8. Concomitant use within 14 days prior to commencement of study treatment of any investigational agent
* 9. Uncontrolled abnormalities of serum potassium, sodium, calcium (corrected) phosphate or magnesium levels
* 10. Pregnant or lactating women. Effective non-hormonal contraception is mandatory for all patients of reproductive potential
* 11. Evidence of ovarian activity
* 12. Prior eribulin therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kenny, Principal Investigator — Consultant Medical Oncologist
Locations (1):
- Charing Cross Hopsital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not currently planned in the protocol.

REFERENCES:
- [Derived] Allsopp RC, Guo Q, Page K, Bhagani S, Kasim A, Badman P, Kenny L, Stebbing J, Shaw JA. Circulating tumour DNA dynamics during alternating chemotherapy and hormonal therapy in metastatic breast cancer: the ALERT study. Breast Cancer Res Treat. 2024 Jul;206(2):377-385. doi: 10.1007/s10549-024-07316-8. Epub 2024 Apr 6. PMID 38581534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a pilot of proof study recruiting 8 breast cancer patients over a 2 year period from the Charing Cross Hospital, London. The last patient completed in July 2018.
Pre-assignment Details: Of the 58 patients screened, during the period between February 2016 and July 2018, 13 patients were consented to the study; and upon screening, 8 were recruited to receive study treatment, eribulin1.23mg/m2 on day 1 and day 8 of 21 day cycles, alternated with an aromatase inhibitor (AI), orally once daily for 9 weeks.
Groups:
- Single Arm Study: 3 x 3 weekly cycles at the recommended dose of eribulin as the ready to use solution, 1.23 mg/m2, administered intravenously over 2-5 minutes on days 1 and 8 of every 21 day cycle. This was then followed by 9 weeks of an Aromatase Inhibitor (AI) treatment (either letrozole, exemestane or anastrozole), followed again by 3 x 3 weekly cycles of eribulin and 9 weeks AI treatment. Patients remained on treatment for up to 9 months, or until disease progression or unacceptable toxicities, whichever was sooner.
Period: Overall Study
Arm/Group | Single Arm Study
Started | 8
Completed | 6
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Patient Non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Study
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [48 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 6
  Ethnicity: Middle Eastern | 1
  Ethnicity: Turkish | 1
  Ethnicity: Mixed | 0
  Ethnicity: Asian | 0
  Ethnicity: Black | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Criteria:
  0 - Fully active, able to carry on all pre-disease activities without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work
  2. - Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. - Capable of only limited self-care, confined to bed or chair 50% or more of waking hours
  4. - Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair
  5. - Death
  Participants
    ECOG Performamce Status 0 | 4
    ECOG Performamce Status 1 | 4
    ECOG Performamce Status 2 | 0
    ECOG Performamce Status 3 | 0
    ECOG Performamce Status 4 | 0
    ECOG Performamce Status 5 | 0
Smoking Status [Count of Participants; unit: Participants]
  Never | 3
  Former | 3
  Current | 1
  No Information | 1
Tumour Type [Count of Participants; unit: Participants]
  Invasive Ducal Carcinoma | 8
  Other Tumour type | 0
Oestrogen Receptor (ER) Status Assessment Method [Count of Participants; unit: Participants] — Hormonal receptors status can be assessed by different methods. Allred scoring method looks at the proportion of positive cells as well as the staining intensity. Other methods report the percentage of positive cells in staining or whether positive or negative.
  Participants
    Allred | 3
    Other | 5
Progesterone Receptors (PgR) Status [Count of Participants; unit: Participants]
  Positive | 7
  Negative | 0
  Unknown | 1
Human Epidermal Growth Factor Receptor 2 (HER2) Status [Count of Participants; unit: Participants] — The IHC test (ImmunoHistoChemistry) uses a chemical dye to stain the HER2 proteins. The IHC gives a score of 0 to 3+ that measures the amount of HER2 proteins on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+, it's considered HER2-negative. If the score is 2+, it's considered borderline. A score of 3+ is considered HER2-positive. If the IHC test results are borderline, it's likely that a FISH test will be done on a sample of the cancer tissue to determine if the cancer is HER2-positive.
  Participants
    Zero | 5
    1+ | 1
    2+ | 0
    3+ | 0
    Not measured | 2
Primary Tumour Stage [Count of Participants; unit: Participants] — Staging is according to the TNM system: Stage 0 (non-invasive), Stage IA, Stage IB, Stage IIA, Stage IIB, Stage IIIA, Stage IIIB, Stage IIIC, Stage IV (worse category).
  Participants
    Stage I | 1
    Stage IIA | 1
    Stage IIIA | 1
    Stage IIIC | 1
    No information | 4
Primary Tumour Grade [Count of Participants; unit: Participants] — The following grades being increasingly malignant over a range of 1 to 4 were adopted:
  G1 Well differentiated (Low grade); G2 Moderately differentiated (Intermediate grade); G3 Poorly differentiated (High grade); G4 Undifferentiated (High grade)
  Participants
    Grade 1 | 1
    Grade 2 | 5
    Grade 3 | 2
Prior Chemotherapy [Count of Participants; unit: Participants]
  Yes | 8
  No | 0
Prior Radiotherapy [Count of Participants; unit: Participants]
  Yes | 8
  No | 0
Prior Surgery [Count of Participants; unit: Participants]
  Yes | 8
  No | 0
Prior Endocrine Therapy [Number; unit: participants]
  Tamoxifen | 8
  Exemestane | 5
  Letrozole | 3
  Anastrozole | 5
Body Mass Index [Median (Full Range); unit: kg/m^2] | 26.5 [20.3 to 31.6]
Primary Tumour Size [Median (Full Range); unit: millimeteres (mm)] | 28 [25 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Estimated Kaplan-Meier Progression Free Survival as Assessed by RECIST v1.1
Description: Estimated Kaplan-Meier Progression free survival (PFS) to be defined as time from study entry to first evidence of disease progression or death due to any cause, as assessed by RECIST v1.0.
Time Frame: Fixed timepoints - 3, 6 and 9 months
Population: PFS was measured at fixed time points of 3, 6 and 9 months, as estimated by the Kaplan-Meier curve. The median PFS at the end of the study was 235 days. PFS could not be calculated at 3 months, as no patient experienced disease progression at follow-up.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Single Arm Study
Number analyzed (Participants) | 8
Days
  3 months | NA [NA to NA] — PFS could not be calculated at 3 months, as no patient experienced disease progression at follow-up.
  6 months | 202 [NA to NA] — A valid confidence interval cannot be accurately calculated for the PFS at 6 months, as only one patient experienced disease progression at follow-up and the given sample size (n=8) is small.
  9 months | 235 [NA to NA] — A valid confidence interval cannot be accurately calculated for the PFS at 9 months, as only three patients experienced disease progression at follow-up and the given sample size (n=8) is small.

2. Secondary Outcome: Clinical Benefit Rate as Assessed by RECIST v1.1
Description: Clinical benefit rate (CBR), defined as the proportion of patients whose best overall response according to Response Evaluation Criteria in Solid Tumours (RECIST), v1.0 is either a complete response, partial response or stable disease for a least 6 months.
Time Frame: To be assessed at 3, 6 and 9 months.
Population: Only 6 patients had at least one tumour assessment during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Study
Number analyzed (Participants) | 6
Participants
  Complete Response | 0
  Partial response | 3
  Stable Disease | 3

3. Secondary Outcome: Safety and Tolerability
Description: Safety and Tolerability were assessed by adverse events (AEs) and serious adverse events (SAEs) according the Common Terminology Criteria for Adverse Event (NCI-CTCAE) v4.03.
Time Frame: Collected form consent to follow-up
Population: AEs and SAEs were collected for all 8 subjects who received at least one dose of study treatment
Measure: Number; unit: Events
Units Other Than Participants: Events
Arm/Group | Single Arm Study
Number analyzed (Participants) | 8
Number analyzed (Events) | 129
Events
  Mild | 71
  Moderate | 39
  Severe | 17
  Life Threatening or disabling | 2
  Death | 0

ADVERSE EVENTS:
Time Frame: Collected from consent to follow-up for all subjects who receive at least one dose of study treatment, 9 months.
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 5/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=8)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) — Patient attended chemo day unit for day 8 eribulin. Routine blood taken prior.; adjusted calcium = 2.96. Patient feeling well within self - no new symptoms/AEs. ECG recorded: normal. IV fluid begun and kept in progress overnight.
Neutopenic Sepsis (Infections and infestations) | 2 (2)
Mucositis (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Patient attended A&E with severe shortness of breath, as hospitalised and treated. Doctors decided to keep the patient longer to have her chest drained before discharging her. Chemotherapy was delayed 1 week to allow the patient to recover.
Respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ischaemia cerebrovascular (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Study (N=8)
Flushing (Vascular disorders) | 2 (2)
Fatigue (General disorders) | 5 (6)
Influenza like illness (General disorders) | 1 (1)
Mucosal inflammation gg (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 3 (4)
Peripheral swelling (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2)
Aspartate aminotransferase (Investigations) | 2 (2)
Blood alkaline phosphatase (Investigations) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Grip strength decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ageusia (Nervous system disorders) | 2 (2)
Diziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 4 (4)
Paraesthesia (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Heartburn/burping (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Teeth and gum darkening (Gastrointestinal disorders) | 1 (1)
Teeth and gum thinning (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Ear infection (Infections and infestations) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 2 (2)
Oral herpes (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT02681523/Prot_SAP_000.pdf